CLINICAL TRIAL: NCT05038033
Title: Addressing Anxiety and Stress for Healthier Eating in Teens
Acronym: ASSET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Metis Foundation (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USUHS.2020-048
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Overweight; Anxiety; Mental Disorders; Body Weight; Eating Behavior; Feeding and Eating Disorders
Keywords: Obesity; Overweight; Anxiety; Adolescent; Prevention; Interpersonal Psychotherapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Obesity; Overweight; Anxiety Disorders; Mental Disorders; Body Weight; Feeding Behavior; Feeding and Eating Disorders | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two treatment arms and two intervention cohorts across two sites.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpersonal Psychotherapy (IPT) (Experimental): Interpersonal Psychotherapy program adapted for the prevention of excessive weight gain. Involves one initial 1.5-hour individual session, and 12 weekly 90-minute group sessions.
  Interventions: Behavioral: Interpersonal Psychotherapy (IPT)
- Cognitive-Behavioral Therapy (CBT) (Active Comparator): The CBT program will match the delivery format and dose of the IPT program. There will be one initial 1.5-hour individual session, and 12 weekly 90-minute group sessions.
  Interventions: Behavioral: Cognitive Behavioral Theory (CBT)

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy (IPT) — The IPT group sessions follow three phases (initial, middle, and termination) and use the interpersonal inventory to identify interpersonal problems that might be contributing to or exacerbating disinhibited eating and anxiety symptoms. A framework of common problem areas is used to teach interpersonal problem-solving and communication skills and educate youth about risk factors and warning signs for excessive weight gain, such as eating in response to negative affect as opposed to hunger, or feeling a sense of loss-of-control while eating. IPT focuses on psychoeducation and general skill-building that can be applied to different relationships within the framework of four interpersonal problem areas: interpersonal role disputes, role transitions, interpersonal deficits, and grief.
  Arms: Interpersonal Psychotherapy (IPT)
Behavioral: Cognitive Behavioral Theory (CBT) — The CBT program will be derived from Coping Cat, a manualized intervention for children and adolescents with elevated symptoms of anxiety. The group intervention builds skills for managing anxiety, in general, but with a focus on how anxiety prompts disinhibited eating, including attention to and restructuring of negative cognitions that perpetuate anxiety and behavioral exposure, rather than avoidance, of anxiety-provoking situations.
  Arms: Cognitive-Behavioral Therapy (CBT)

SUMMARY:
Project ASSET will explore the preliminary efficacy of interpersonal therapy, when compared with cognitive behavioral therapy, for reducing anxiety symptoms, preventing excess weight gain, and reducing cardio-metabolic risk in adolescent girls with above-average weight and elevated anxiety. As a pilot for a larger multi-site study, this trial will also test multi-site feasibility, acceptability, and intervention fidelity.

DETAILED DESCRIPTION:
This study is a randomized controlled trial in which 40 adolescent girls aged 12-17 years-old with weight in the 75th percentile or higher for their age and sex, and elevated anxiety symptoms, will be randomly assigned to an IPT or CBT 12-week group intervention. Approximately 20 adolescent girls will be enrolled at each of two sites: Uniformed Services University (USU) and Colorado State University (CSU). After a screening and baseline assessment, participants will attend an individual meeting with the leaders of their assigned group to learn more about the group process and establish goals. They will then participate in the group program for 12 consecutive weeks. Each group will be led by a PhD-level clinical psychologist and a healthcare trainee. In-person and remote assessments, will be conducted at baseline, in the ~two weeks post-intervention (i.e., 12-week follow-up), and at 1, 2, and 3 years post-intervention. These assessments will consist of body measurements, blood draws for collection markers of metabolic functioning, and surveys and interviews of psychological and social functioning. At baseline, two weeks, and one year post-intervention, participants will also have a week-long period during which they will wear devices collecting activity and physiological data, and complete phone surveys assessing disinhibited eating behaviors, food craving, affect, cognitions, and avoidance behaviors.

ELIGIBILITY:
Participant Inclusion Criteria:

* 12-17-year-old adolescent girls
* BMI ≥ 75th percentile
* Anxiety symptoms: 32 or higher on State Trait Anxiety Inventory for Children-Trait Scale

Participant Exclusion Criteria:

* Any medical condition (as well as pregnancy or breastfeeding)
* Individuals who have any DSM psychiatric disorder that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study
* Medication impacting mood or weight
* Psychotherapy

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Intervention Fidelity and Acceptability | Entirety of the Study
  Feasibility: Fidelity ratings of facilitators' competence/adherence in administration of IPT and CBT; CONSORT tracking of recruitment, recruitment rate and percentage of eligible adolescents who enroll as recorded by study coordinators; median sessions attended and home practice completion, as recorded by facilitators; CONSORT tracking of follow-up retention as recorded by study coordinators; and completeness of data collection.
  Acceptability: Adolescent self-reports on program and monitor acceptability questionnaires

SECONDARY OUTCOMES:
Presence of Disinhibited Eating | Post-Treatment
  Eating Disorder Examination Interview- overeating section will be administered to assess for the presence of overeating with and without loss of control.
Mood/Anxiety, Eating, And Social Functioning | Post Treatment
  Adolescent self-reports on mood and eating as well as psychological distress via questionnaire, interview, and smartphone surveys.
  Assesed through completion of surveys: Center For Epidemiologic Studies - Depression Scale (CES-D), Social Phobia And Anxiety Inventory For Children (SPAI-C), Emotional Eating Scale - Children, Social Adjustment Scale-self Report, Difficulties In Emotion Regulation Scale-short Form, Conflict Behavior Questionnaire, Network Of Relationships Inventory-short Form, Children's Automatic Thoughts Scale (CATS-N/P), Anxiety Control Questionnaire For Children (ACQ-C), The Self-efficacy Questionnaire For Children (SEQ-C), Children's Coping Strategies Checklist - Revised (CCSC-R1), Positive And Negative Affect Schedule - Child Form (PANAS-C).
Participant Height, Weight, and Blood Pressure | Post Treatment
  Weight will be measured via scale and height via stadiometer. This will be used to calculate BMI percentile. Blood pressure assessed via digital blood pressure monitor.
Body Composition Measurement | Post treatment
  Assessed using air displacement plethysmography (Bod Pod).
Collection of Metabolic Markers | Post Treatment
  Blood will be drawn in a fasted state to measure glucose, insulin, and lipids.
Parental report of eating behaviors | Post Treatment
  Parents/guardians will be asked to complete Eating in the Absence of Hunger Questionnaire for Children - Parent Report (EAH-C Parent).
Cardiometabolic Functioning | Post Treatment
  Measured by blood draw, continuous glucose monitoring, and heart rate, sleep and activity via Carnation Ambulatory Monitor.
Movement and Activity | Post Treatment
  Measured by ActivPal monitoring device

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Colorado State University, Fort Collins, Colorado
  - Uniformed Services University, Bethesda, Maryland